CLINICAL TRIAL: NCT03247751
Title: Rotational Stability of the Blue Light-absorbing Hydrophobic Acrylic Posterior Chamber Single Piece Intraocular Lens
Brief Title: Evaluation of the Rotational Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPF001C
Record Dates: First submitted 2017-06-16; First posted 2017-08-14 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one group (Experimental): one group receiving NIDEK intraocular lens
  Interventions: Device: intraocular lens

INTERVENTIONS:
Device: intraocular lens — Implant NIDEK intraocular lens after cataract surgery

SUMMARY:
To evaluate rotational stability of the investigational device implanted after cataract surgery.

DETAILED DESCRIPTION:
The primary endpoint is angle of intraocular lens rotation between the day of surgery and postoperative 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years or older
* Subject who diagnosed unilateral or bilateral age-related cataract.
* Potential postoperative BCVA of 0.2 log MAR (0.63) or better.
* Calculated IOL power in within the range of investigational IOL.
* Subject is able to understand, agree and sign the informed consent statement.
* Subject is able and willing to comply with the postoperative follow-up examination schedule.

Exclusion Criteria:

* Uncontrolled systemic or ocular disease.
* Extremely shallow anterior chamber.
* Previous intraocular and corneal surgery.
* Traumatic cataract.
* Pregnancy or lactation.
* Concurrent participation in another drug and device clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The intraocular lens rotation | postoperative 6 months
  The angle of the intraocular rotation.

SECONDARY OUTCOMES:
visual acuity | postoperative 6 months
  Distance BCVA
Adverse event | postoperative 6 months
  severity and causal relationship

IPD SHARING:
Plan to Share IPD: No